CLINICAL TRIAL: NCT00346398
Title: A Phase II Multicenter, Controlled, Double-Blind Study Using Immunoprophylaxis in the Primary Prevention of Allergic Disease (ITN025AD)
Brief Title: Promoting Tolerance to Common Allergens in High-Risk Children: Global Prevention of Asthma in Children (GPAC) Study
Acronym: GPAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DAIT ITN025AD
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Asthma; Allergic Sensitization
Keywords: asthma; allergen; allergic disease; allergen immunotherapy; allergic sensitization; atopic dermatitis; eczema; food allergy; oral mucosal immunoprophylaxis (OMIP)
MeSH Terms: conditions — Asthma; Dermatitis, Atopic; Eczema; Food Hypersensitivity | interventions — Desensitization, Immunologic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral mucosal immunoprophylaxis (OMIP) (Experimental): Participants are administered oral mucosal immunoprophylaxis (OMIP) daily for 12 months.
  Interventions: Biological: Oral mucosal immunoprophylaxis (OMIP)
- Placebo (Placebo Comparator): Participants are administered, via the same route as the experimental group, an oral placebo solution daily for 12 months.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Oral mucosal immunoprophylaxis (OMIP) — OMIP consists of a mixture of allergen extracts including 0.2 milliliters (mL) timothy grass, 0.2 mL cat, and 0.2 mL house dust mite for a total daily dose of 0.6 mL.
  Other Names: Allergen immunotherapy
  Arms: Oral mucosal immunoprophylaxis (OMIP)
Biological: Placebo — The placebo consists of three 0.2 mL vials of solution mixed together for a total daily dose of 0.6 mL.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether early childhood exposure to common allergens (substances that can trigger allergies and asthma) can prevent the development of asthma in children at high risk for developing the disease.

DETAILED DESCRIPTION:
Researchers suspect that allergies to common inhaled allergens (such as house dust mite, cat dander, and grass pollens) are a major cause of childhood asthma. Recent evidence suggests that if allergies to inhaled allergens are prevented, this can cause changes in the immune system that may inhibit the development of asthma. Although strategies to prevent allergies generally focus on avoiding the allergen, complete avoidance of the common allergens linked to asthma would require extreme measures and is impractical.

Oral mucosal immunoprophylaxis (OMIP) therapy is an allergy treatment that can induce long-lasting immune tolerance in people already suffering from allergies. By exposing the patient to small, repeated, but increasing doses of the problem allergen over a long period of time, the patient's immune system is eventually desensitized to that particular allergen. OMIP therapy has been shown to be safe in children as young as 2 years old. This study will evaluate if OMIP therapy against common inhaled allergens is safe and effective in preventing the development of asthma in children at high risk for developing the disease. Children enrolled in this study have been diagnosed with eczema or food allergies and have a family history of eczema, allergic rhinitis, or asthma.

There are two groups in this study. The experimental arm participants will receive OMIP therapy (a mixture of house dust mite, cat, and timothy grass allergens) as daily oral drops under the tongue for 1 year; Placebo arm participants will receive an allergen free placebo solution. Participants will be followed for an additional 3 years to see whether they develop allergies or asthma and to determine how OMIP affects their immune system's response to allergens. There will be 5 study visits in the first year and 6 visits over the next 3 years. At all visits, participants will be assessed for allergy/asthma symptoms, will be asked to complete questionnaires, and may be asked to provide blood or saliva samples.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with eczema (atopic dermatitis)
* Family history of eczema, allergic rhinitis, or asthma
* Allergy to one or more of the following: egg white, cow's milk, peanut, or soybean
* Weigh at least 9.5 kg (20.9 lbs)
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* Allergy to house dust mite, cat, or timothy grass
* Born prematurely (before 36th week's gestation)
* Previous diagnosis of asthma OR have had 3 or more distinct episodes of wheeze during the first year of life
* Chronic pulmonary disease
* Chronic disease requiring therapy
* Past or current treatment with systemic immunomodulator medication
* Past or current treatment with allergen-specific immunotherapy
* Received 10 or more days of systemic steroids in the 3 months prior to study entry
* Orofacial abnormalities that are likely to interfere with the subject's ability to take study treatment
* Participated in another clinical study within the 3 months prior to study entry

Ages: 12 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2006-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Holt, MD, Principal Investigator — Telethon Institute for Child Health Research; Peter Sly, MD, Study Chair — Telethon Institute for Child Health Research
Locations (3):
- Mount Sinai School of Medicine, New York, New York, United States
- Australia (2):
  - Royal Children's Hospital, Melbourne, Victoria
  - Telethon Institute for Child Health Research, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Data access is provided to the public in: 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools available to researchers; and 2.) TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal that makes data from the consortium's clinical trials publicly available.

REFERENCES:
- [Background] Mascarell L, Van Overtvelt L, Moingeon P. Novel ways for immune intervention in immunotherapy: mucosal allergy vaccines. Immunol Allergy Clin North Am. 2006 May;26(2):283-306, vii-viii. doi: 10.1016/j.iac.2006.02.009. PMID 16701145
- [Background] Nelson HS. Advances in upper airway diseases and allergen immunotherapy. J Allergy Clin Immunol. 2006 May;117(5):1047-53. doi: 10.1016/j.jaci.2005.12.1306. Epub 2006 Mar 6. PMID 16675331
- [Result] Holt PG, Sly PD, Sampson HA, Robinson P, Loh R, Lowenstein H, Calatroni A, Sayre P. Prophylactic use of sublingual allergen immunotherapy in high-risk children: a pilot study. J Allergy Clin Immunol. 2013 Oct;132(4):991-3.e1. doi: 10.1016/j.jaci.2013.04.049. Epub 2013 Jun 12. No abstract available. PMID 23768574
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org
- Available data/document: Individual Participant Data Set: SDY545 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY545 — ImmPort study identifier is SDY545.
- Available data/document: Study summary, -design with synopsis, -adverse events, -assessment, -medications, -demographics, -lab tests, -files, et al.: SDY545 — http://www.itntrialshare.org/project/Studies/ITN025ADPUBLIC/Study%20Data/begin.view? — ImmPort study identifier is SDY545.
- Available data/document: Individual Participant Data Set: ITN025AD — http://www.itntrialshare.org/project/Studies/ITN025ADPUBLIC/Study%20Data/begin.view? — TrialShare is the ITN clinical trials research portal available to the public.
- Available data/document: Study overview with synopsis, -navigator, -schedule of events, -data and reports, biospecimens and availability.: ITN025AD — http://www.itntrialshare.org/project/Studies/ITN025ADPUBLIC/Study%20Data/begin.view? — TrialShare study identifier is ITN025AD.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred between June 2006 and July 2007 at 2 sites in Australia and 1 site in the United States
Pre-assignment Details: At a screening visit, subjects underwent procedures to establish that all inclusion criteria were met and none of the exclusion criteria were met. All guardians provided written informed consent
Groups:
- OMIP With Timothy Grass, Cat and House Dust Mite Allergens: Participants were administered oral mucosal immunoprophylaxis (OMIP) daily for 12 months. OMIP consisted of a mixture of allergen extracts including 0.2 milliliters (mL) timothy grass, 0.2 mL cat, and 0.2 mL house dust mite for a total daily dose of 0.6 mL. After 12 months, treatment stopped and participants were tested 3 years after end of treatment for development of allergic sensitization and asthma.
- Placebo: Participants were administered via the same route as the experimental group an oral placebo solution daily for 12 months. The placebo consisted of three 0.2 mL vials of solution mixed together for a total daily dose of 0.6 mL. After 12 months, treatment stopped and participants were tested 3 years after end of treatment for development of allergic sensitization and asthma.
Period: Overall Study
Arm/Group | OMIP With Timothy Grass, Cat and House Dust Mite Allergens | Placebo
Started | 25 | 26
Completed | 22 | 24
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OMIP With Timothy Grass, Cat and House Dust Mite Allergens | Placebo | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Customized [Number; unit: participants]
  Aged 12-17 Months | 6 | 6 | 12
  Aged 18-23 Months | 16 | 12 | 28
  Aged 24-30 Months | 3 | 8 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 12 | 14 | 26
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8
  Australia | 21 | 22 | 43
Severity of Atopic Dermatitis (AD) Using SCORAD Index [Mean (Standard Deviation); unit: Units on a Scale] — Scoring of Atopic Dermatitis (SCORAD) disease-severity scale measures intensity of erythema, edema/papulation, oozing/crusts, excoriations, lichenification and dryness, each on a scale from 0-3 for a maximum total of 18 points. This score is multiplied by 3.5 and added to 1/5 of the affected percent body surface area. The final score is added to the score from a 0-10 point pruritus visual analog scale (VAS) and a 0-10 point loss of sleep VAS. Summary: SCORAD (0-103)=extent (0-100)/5+intensity (0-18)x3.5 + pruritus and sleep (0-20).Interpretation: SCORAD (0 (no disease) to 103 (most severe)).
  Units on a Scale | 13.3 (8.5) | 11.4 (9.1) | 12.3 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Allergic Sensitization at Month 36 Status Post Treatment Completion
Description: Allergic sensitization is defined as a positive serum allergen specific Immunoglobulin E (IgE) CAP test[1] or a positive allergy skin prick test[2]. Not experiencing allergic sensitization is the better outcome for this measure.
  1. A positive serum allergen specific IgE CAP (ImmunoCAP) test result is defined by a result >= 0.35 kU/L. Higher scores indicate greater allergic sensitization.
  2. A positive skin prick test is defined as a wheal diameter that is 3 mm larger than that produced by a negative control. Higher wheal sizes indicate greater allergic reaction or sensitization.
Time Frame: Three years (36 months) after Treatment Completion
Population: Intent-to-treat minus one participant in placebo group who had a sibling in trial
Measure: Number; unit: participants
Arm/Group | OMIP With Timothy Grass, Cat and House Dust Mite Allergens | Placebo
Number analyzed (Participants) | 25 | 25
participants | 22 | 19
Statistical Analysis 1: Comparison: OMIP With Timothy Grass, Cat and House Dust Mite Allergens vs Placebo; Participants who drop out (have missing efficacy endpoints) are considered treatment failures; Test type: Superiority or Other; p = 0.28, Chi-squared — Odds Ratios are calculated using a logistic regression with a Wald chi square test. Experimental group participants had a higher proportion of allergic sensitization than participants who received placebo; Odds Ratio (OR) = 2.3, 95% CI 2-sided [0.5 to 10.5]

2. Secondary Outcome: Number of Participants With Current Asthma at Month 36 Status Post Treatment Completion
Description: Participants who currently have asthma three years after end of treatment. Asthma is defined as three distinct episodes of wheeze after the first year of life, each of which lasts 3 or more consecutive days and occurs in a clinical setting where asthma is likely and other likely conditions have been excluded. Episodes must be separated by at least 7 days without wheeze. Current asthma is defined as a diagnosis of asthma and at least one episode of wheeze lasting 3 or more consecutive days in the past 12 months.
Time Frame: Three years (36 months) after Treatment Completion
Population: Intent-to-treat minus one participant in placebo group who had a sibling in trial
Measure: Number; unit: participants
Arm/Group | OMIP With Timothy Grass, Cat and House Dust Mite Allergens | Placebo
Number analyzed (Participants) | 25 | 25
participants | 4 | 4
Statistical Analysis 1: Comparison: OMIP With Timothy Grass, Cat and House Dust Mite Allergens vs Placebo; Participants who drop out (have missing efficacy endpoints) are considered treatment failures; Test type: Superiority or Other; p = 0.85, Chi-squared — Odds Ratios are calculated using unadjusted exact logistic regression with mid p-value to adjust for the discreteness of the distribution; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.2 to 6.1]

3. Secondary Outcome: Time to First Onset of Asthma
Description: Time to first onset of asthma is the time from the day a participant is randomized and initiates study treatment to the diagnosis of the first of three episodes of asthma. Asthma is defined as three distinct episodes of wheeze after the first year of life, each of which lasts 3 or more consecutive days and occurs in a clinical setting where asthma is likely and other likely conditions have been excluded. Episodes must be separated by at least 7 days without wheeze.
Time Frame: From Treatment Initiation to Month 36 Status Post Treatment Completion
Population: Intent-to-treat minus one participant in placebo group who had a sibling in trial
Measure: Mean (Standard Error); unit: Months
Arm/Group | OMIP With Timothy Grass, Cat and House Dust Mite Allergens | Placebo
Number analyzed (Participants) | 25 | 25
Months | 31.0 (1.9) | 38.3 (2.1)
Statistical Analysis 1: Comparison: OMIP With Timothy Grass, Cat and House Dust Mite Allergens vs Placebo; Test type: Superiority or Other; p = 0.28, Regression, Logistic — P-value is calculated using a log-rank test; Hazard Ratio (HR) = 1.8, 95% CI 2-sided [0.6 to 5.6] — Hazard ratio and 95% confidence intervals are calculated using an unadjusted Cox regression

ADVERSE EVENTS:
Time Frame: Start of study through three years post-treatment (up to four years total)
Description: This study graded the severity of adverse events experienced by the study participant according to criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.0 (June 10, 2003). One participant in the placebo group is included in adverse event reports, but excluded from further analysis.
Arm/Group | OMIP With Timothy Grass, Cat and House Dust Mite Allergens | Placebo
Serious Adverse Events (participants affected / at risk) | 8/25 | 7/26
Other Adverse Events (participants affected / at risk) | 25/25 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMIP With Timothy Grass, Cat and House Dust Mite Allergens (N=25) | Placebo (N=26)
Conductive deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Breathing-related sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMIP With Timothy Grass, Cat and House Dust Mite Allergens (N=25) | Placebo (N=26)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 5 (6)
Conjunctivitis (Eye disorders) | 8 (23) | 14 (20)
Conjunctivitis allergic (Eye disorders) | 5 (5) | 3 (3)
Eye pruritus (Eye disorders) | 3 (4) | 5 (12)
Lacrimation increased (Eye disorders) | 6 (11) | 8 (18)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 1 (2)
Constipation (Gastrointestinal disorders) | 4 (6) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 17 (32) | 21 (57)
Oral pruritus (Gastrointestinal disorders) | 2 (7) | 1 (1)
Teething (Gastrointestinal disorders) | 8 (10) | 8 (22)
Vomiting (Gastrointestinal disorders) | 15 (34) | 18 (52)
Pyrexia (General disorders) | 18 (60) | 19 (51)
Allergy to animal (Immune system disorders) | 2 (2) | 3 (11)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 1 (1)
Food allergy (Immune system disorders) | 9 (35) | 8 (20)
Hypersensitivity (Immune system disorders) | 7 (28) | 6 (14)
Seasonal allergy (Immune system disorders) | 4 (12) | 4 (5)
Bronchitis (Infections and infestations) | 3 (3) | 1 (2)
Croup infectious (Infections and infestations) | 1 (4) | 2 (2)
Ear infection (Infections and infestations) | 10 (15) | 6 (17)
Gastroenteritis (Infections and infestations) | 13 (30) | 12 (26)
Lower respiratory tract infection (Infections and infestations) | 3 (9) | 4 (7)
Nasopharyngitis (Infections and infestations) | 21 (141) | 23 (145)
Otitis media (Infections and infestations) | 4 (14) | 3 (4)
Otitis media acute (Infections and infestations) | 3 (5) | 4 (7)
Pharyngitis (Infections and infestations) | 1 (1) | 3 (4)
Respiratory tract infection viral (Infections and infestations) | 3 (4) | 2 (7)
Rhinitis (Infections and infestations) | 7 (18) | 5 (9)
Tonsillitis (Infections and infestations) | 7 (11) | 7 (17)
Upper respiratory tract infection (Infections and infestations) | 22 (192) | 24 (184)
Urinary tract infection (Infections and infestations) | 3 (5) | 3 (6)
Varicella (Infections and infestations) | 2 (2) | 6 (6)
Viral infection (Infections and infestations) | 12 (36) | 10 (26)
Arthropod bite (Injury, poisoning and procedural complications) | 4 (6) | 3 (5)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Febrile convulsion (Nervous system disorders) | 2 (5) | 1 (2)
Headache (Nervous system disorders) | 4 (5) | 4 (11)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (25) | 4 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (111) | 20 (83)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (14) | 3 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 (27) | 12 (48)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 2 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 20 (82) | 20 (99)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 11 (33) | 8 (20)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (7) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 11 (62) | 10 (31)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 11 (25) | 7 (12)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (12) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 8 (20) | 6 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 9 (28) | 6 (9)

LIMITATIONS AND CAVEATS:
One participant in the placebo group could not be included in intent-to-treat analyses because a sibling was also in the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No